CLINICAL TRIAL: NCT06742814
Title: Effects of Stress Ball Use for Patients Undergoing Local Anesthesia in Ambulatory Surgery: A Randomized Controlled Trial
Brief Title: Effects of Stress Ball Use for Patients Undergoing Local Anesthesia in Ambulatory Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202408018RIND
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-09

CONDITIONS: Anxiety
Keywords: anxiety; stress ball; ambulatory surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): usal nursing care
- intervation group (Experimental): stress ball
  Interventions: Device: stress ball

INTERVENTIONS:
Device: stress ball — Stress ball: It is a ball with moderate hardness and softness, about 6 cm, which can be held and pressed by hand.
  Arms: intervation group

SUMMARY:
Preoperative anxiety begins from the decision-making of surgery to entering the operating room and may intensify as the surgery date approaches. Anxiety not only causes physiological effects but also psychological impacts, leading to negative outcomes for postoperative recovery. Ambulatory surgeries often employ local anesthesia, where patients remain conscious during the procedure, potentially causing specific anxieties and fears. The use of a stress ball is a non-pharmacological method that effectively distracts individuals consciously focusing on stimuli. This study is expected to be a randomized controlled trial, using convenience sampling to select patients receiving local anesthesia. They will be divided into two groups through computer-generated random number sequences: the stress ball group and the control group. The research aims to alleviate anxiety and pain levels in outpatient surgery patients receiving local anesthesia, with the goal of improving patients' postoperative mental health and quality of care.

ELIGIBILITY:
Inclusion Criteria:

- 1. Those who are over 18 years old, have clear consciousness and can communicate in Chinese and Taiwanese Hakka.

2. Patients undergoing outpatient surgery under local anesthesia.

Exclusion Criteria:

* Unable to cooperate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 3 minutes
  It is a physiological monitoring indicator. When the human body receives internal and external environmental stimuli, the autonomic nervous system regulates the heart rhythm to perform a series of responses to the stimulus source (Huang et al., 2008). Heart Rate Variability (HRV) is an objective physiological indicator that can be used An assessment tool for anxiety status during surgery (Correa et al., 2021; Tang et al., 2006).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory, S-TAI | 5 - 10 minutes
  It is based on the individual's feelings in a specific situation.
Visual Analogue Scale | 3 minutes
  Measure the patient's pain level using VAS 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Ling Chang, Study Chair — NTUH Hsin-Chu Branch

IPD SHARING:
Plan to Share IPD: No
1. Assessing changes in patient anxiety and pain during outpatient surgery
  2. To explore the impact of pressure balls on patients' anxiety and pain during outpatient surgery

REFERENCES:
- [Result] Boonstra AM, Schiphorst Preuper HR, Balk GA, Stewart RE. Cut-off points for mild, moderate, and severe pain on the visual analogue scale for pain in patients with chronic musculoskeletal pain. Pain. 2014 Dec;155(12):2545-2550. doi: 10.1016/j.pain.2014.09.014. Epub 2014 Sep 17. PMID 25239073
- [Result] Haugen AS, Eide GE, Olsen MV, Haukeland B, Remme AR, Wahl AK. Anxiety in the operating theatre: a study of frequency and environmental impact in patients having local, plexus or regional anaesthesia. J Clin Nurs. 2009 Aug;18(16):2301-10. doi: 10.1111/j.1365-2702.2009.02792.x. PMID 19583663
- [Result] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687
- [Result] Karatas TC, Gezginci E. The Effect of Using a Stress Ball During Endoscopy on Pain, Anxiety, and Satisfaction: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):309-317. doi: 10.1097/SGA.0000000000000739. Epub 2023 May 17. PMID 37199436
- [Result] Klopfenstein CE, Forster A, Van Gessel E. Anesthetic assessment in an outpatient consultation clinic reduces preoperative anxiety. Can J Anaesth. 2000 Jun;47(6):511-5. doi: 10.1007/BF03018941. PMID 10875713
- [Result] Lee A, Chui PT, Gin T. Educating patients about anesthesia: a systematic review of randomized controlled trials of media-based interventions. Anesth Analg. 2003 May;96(5):1424-1431. doi: 10.1213/01.ANE.0000055806.93400.93. PMID 12707146
- [Result] Maheshwari D, Ismail S. Preoperative anxiety in patients selecting either general or regional anesthesia for elective cesarean section. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):196-200. doi: 10.4103/0970-9185.155148. PMID 25948900
- [Result] Myles PS, Urquhart N. The linearity of the visual analogue scale in patients with severe acute pain. Anaesth Intensive Care. 2005 Feb;33(1):54-8. doi: 10.1177/0310057X0503300108. PMID 15957691
- [Result] Myles PS, Myles DB, Galagher W, Boyd D, Chew C, MacDonald N, Dennis A. Measuring acute postoperative pain using the visual analog scale: the minimal clinically important difference and patient acceptable symptom state. Br J Anaesth. 2017 Mar 1;118(3):424-429. doi: 10.1093/bja/aew466. PMID 28186223
- [Result] Salamon E, Kim M, Beaulieu J, Stefano GB. Sound therapy induced relaxation: down regulating stress processes and pathologies. Med Sci Monit. 2003 May;9(5):RA96-RA101. PMID 12761468
- [Result] Soltani P, Moaddabi A, Koochek Dezfuli M, Ebrahimikiyasari S, Hosseinnataj A, Rengo S, Tavakoli Tafti K, Spagnuolo G. Evaluating the effect of using anti-stress balls as a distraction technique in reducing pain during inferior alveolar nerve block injection: a randomized clinical trial. Clin Oral Investig. 2023 Aug;27(8):4653-4658. doi: 10.1007/s00784-023-05091-2. Epub 2023 Jun 17. PMID 37328611
- [Result] Sriramka B, Mallik D, Singh J, Khetan M. Effect of hand-holding and conversation alone or with midazolam premedication on preoperative anxiety in adult patients-A randomised controlled trial. Indian J Anaesth. 2021 Feb;65(2):128-132. doi: 10.4103/ija.IJA_705_20. Epub 2021 Feb 10. PMID 33776087
- [Result] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- See also: Global prevalence and determinants of preoperative anxiety among surgical patients: A systematic review and meta-analysis — https://doi.org/10.1016/j.ijso.2020.05.010
- See also: Influence of anxiety on the heart rate variability of patients in preoperative orthopedic surgery — https://doi.org/10.33448/rsd-v10i8.17237